CLINICAL TRIAL: NCT00479687
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled Trial of SUPARTZ (Sodium Hyaluronate) for the Treatment of Chronic Shoulder Pain
Brief Title: SUPARTZ Versus Placebo in Osteoarthritis of the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHO-0106
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: Osteoarthritis; Shoulder; Hyaluronic Acid (HA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supartz (Active Comparator): SUPARTZ® 3 injections over 2 weeks
  Interventions: Device: SUPARTZ®
- Phosphate Buffered Saline (Placebo Comparator): Phosphate Buffered Saline 3 injections over 2 weeks
  Interventions: Device: Phosphate Buffered Saline

INTERVENTIONS:
Device: SUPARTZ® — Three Supartz injections over 2 weeks into the glenohumeral joint space.
  Arms: Supartz
Device: Phosphate Buffered Saline — Three phosphate buffered saline injections over 2 weeks into the glenohumeral joint space.
  Other Names: Saline
  Arms: Phosphate Buffered Saline

SUMMARY:
This clinical trial is to determine the safety and effectiveness of three injections of SUPARTZ (sodium hyaluronate) compared with phosphate buffered saline (PBS) for the treatment of glenohumeral osteoarthritis of the shoulder. The trial contains two phases. Phase I is 26 weeks, double blinded, and subjects are randomized to either SUPARTZ or PBS treatment. Phase II is 26 weeks (total 52 weeks) and open-label so all subjects will receive SUPARTZ injections only.

DETAILED DESCRIPTION:
Phase 3 Study: Multi-center, randomized, double blinded, two phase study to determine the safety and efficacy of 3 injections of SUPARTZ for Osteoarthritis of the Shoulder

ELIGIBILITY:
Inclusion Criteria:

* Glenohumeral Osteoarthritis (OA) confirmed by radiograph
* Limitation of shoulder motion in at least one direction
* Retained active range of motion of at least 30% in all directions

Exclusion Criteria:

* Full thickness rotator cuff tear or rotator cuff tendinopathy
* Frozen shoulder
* Female who is pregnant or lactating

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sledge, MD, Principal Investigator — Northeast Orthopedics - Unlimited Research; Charles Birbara, MD, Principal Investigator — Clinical Pharmacology Study Group

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph1: Supartz (Double Blind); Ph2: Supartz (Open Label): SUPARTZ® 3 injections over 2 weeks
  SUPARTZ®: Three Supartz injections over 2 weeks into the glenohumeral joint space.
- Ph1: Phosphate Buffered Saline (Double Blind): Phosphate Buffered Saline 3 injections over 2 weeks
  Phosphate Buffered Saline: Three phosphate buffered saline injections over 2 weeks into the glenohumeral joint space.
Period: Ph 1: Blinded, Randomized, Controlled
Arm/Group | Ph1: Supartz (Double Blind) | Ph1: Phosphate Buffered Saline (Double Blind) | Ph2: Supartz (Open Label)
Started | 150 | 150 | 0
Completed | 125 | 131 | 0
Not Completed | 25 | 19 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 5 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 11 | 0
Period: Ph 2: Open Label, Single (Supartz) Arm
Arm/Group | Ph1: Supartz (Double Blind) | Ph1: Phosphate Buffered Saline (Double Blind) | Ph2: Supartz (Open Label)
Started | 0 | 0 | 224 (Four did not continue to Ph2; 224 received at least 1 inj. and 28 received no trt. (only follow-up))
Completed | 0 | 0 | 215
Not Completed | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Double Blind = Intention-to-treat (ITT): all subjects randomized Open Label = Retreatment Subjects, All ITT subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph1: Supartz (Double Blind) | Ph1: Phosphate Buffered Saline (Double Blind) | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 65 | 133
  >=65 years | 82 | 85 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.7) | 65.7 (11.8) | 65.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 75 | 136
  Male | 89 | 75 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 146 | 144 | 290
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 8 | 14
  White | 143 | 140 | 283
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS: 0-100) for Pain on Movement
Description: Visual Analogue Scale (VAS) for pain on (shoulder) movement with a range of 0 to100; where 0=No pain at all and 100=Pain as bad as it can be.
  Q: How bad is the pain in your study shoulder with activity or movement? (For example, when putting on a coat, sleeping on your study shoulder side, combing your hair, reaching a high shelf, etc.)
  Reported is a single Least square mean point estimate over the 7-26 week time interval using the assessments collected at weeks 7, 13, 20, and 26
Time Frame: Ph1: weeks 7 - 26
Population: Glenohumeral Osteoarthritis (GH-OA) Intention-to-Treat (ITT) population includes all randomized subjects who had no clinical diagnosis of concomitant pathologies in the trial shoulder
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ph1: Supartz (Double Blind) | Ph1: Phosphate Buffered Saline (Double Blind)
Number analyzed (Participants) | 133 | 130
units on a scale | 53.7665 (1.7513) | 57.7659 (1.7569)
Statistical Analysis 1: Comparison: Ph1: Supartz (Double Blind) vs Ph1: Phosphate Buffered Saline (Double Blind); Test type: Superiority; p = 0.0380, Mixed Models Analysis — There was a single primary variable and the a-prior threshold for statistical significance was 0.05; mixed effects repeated measure model with baseline VAS, treatment, and week as fixed effects and subject nested within site as a random effect

ADVERSE EVENTS:
Time Frame: 52 weeks: Ph1 (Double Blind) from baseline week 0 to week 26 (26 weeks); Ph2 (Open Label) week 26 to week 52 (26 weeks)
Description: This study had 2 phases. Phase 1 was double blind for 26 weeks. Phase 2 was an open label extension for 26 weeks.
Groups:
- Supartz (Double Blind); Supartz (Open Label): SUPARTZ® 3 injections over 2 weeks
  SUPARTZ®: Three Supartz injections over 2 weeks into the glenohumeral joint space.
- Phosphate Buffered Saline (Double Blind): Phosphate Buffered Saline 3 injections over 2 weeks
  Phosphate Buffered Saline: Three phosphate buffered saline injections over 2 weeks into the glenohumeral joint space.
Arm/Group | Supartz (Double Blind) | Phosphate Buffered Saline (Double Blind) | Supartz (Open Label)
Serious Adverse Events (participants affected / at risk) | 11/150 | 5/150 | 5/224
Other Adverse Events (participants affected / at risk) | 54/150 | 56/150 | 21/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supartz (Double Blind) (N=150) | Phosphate Buffered Saline (Double Blind) (N=150) | Supartz (Open Label) (N=224)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Bone fragmentation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Supartz (Double Blind) (N=150) | Phosphate Buffered Saline (Double Blind) (N=150) | Supartz (Open Label) (N=224)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 46 | 53 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No